CLINICAL TRIAL: NCT00004386
Title: Phase I Pilot Study of Liver-Directed Gene Therapy for Partial Ornithine Transcarbamylase Deficiency
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: Children's National Research Institute (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/12054; CSH-3660
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-01

CONDITIONS: Ornithine Transcarbamylase Deficiency Disease
Keywords: inborn errors of metabolism; rare disease; urea cycle disorder
MeSH Terms: conditions — Ornithine Carbamoyltransferase Deficiency Disease; Metabolism, Inborn Errors; Rare Diseases; Urea Cycle Disorders, Inborn

INTERVENTIONS:
Genetic: recombinant adenovirus containing the ornithine transcarbamylase gene

SUMMARY:
OBJECTIVES:

Evaluate the safety and feasibility of administering recombinant adenovirus containing the ornithine transcarbamylase gene to adults with partial ornithine transcarbamylase deficiency.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This a dose escalation study to estimate the maximum tolerated dose of recombinant adenovirus encoded with the ornithine transcarbamylase gene.

Patients receive a single dose of virus infused into the liver under fluoroscopic guidance. Groups of 3 patients receive successively higher doses of virus; each cohort is observed for safety for 3 weeks before entry of the next group.

Patients are followed weekly for 1 month, then every 3 months until stable.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Confirmed partial ornithine transcarbamylase deficiency Asymptomatic, i.e., at least 1 month since hyperammonemia --Prior/Concurrent Therapy-- Not specified --Patient Characteristics-- No pregnant or nursing women Negative pregnancy test required of fertile women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1995-10

CONTACTS AND LOCATIONS:
Overall Officials: Mark Batshaw, Study Chair — Children's National Research Institute